CLINICAL TRIAL: NCT00180726
Title: Regulation of Inflammatory Mediators in Asthma
Brief Title: Molecular Mechanism of Asthma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NHLI-MB-1
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Asthma
Keywords: asthma, inflammatory, corticosteroid
MeSH Terms: conditions — Asthma | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Blood sampling, Endoscopic Bronchoscopy, Spirometry

SUMMARY:
The aim of this study is to investigate the mechanisms whereby lung function is decreased in asthma and sensitivity to treatment. The hypothesis is that in diseases such as asthma, inflammatory cells (leukocytes) including eosinophils, macrophages and lymphocytes migrate to the lung and release either more or different types of inflammatory mediators and/or receptors compared to subjects without asthma, which are corticoid sensitive or insensitive. The objective of the study is to identify which genes are specifically expressed in important cells in patients with asthma with a view to identify novel targets for drug therapy.

DETAILED DESCRIPTION:
We aim to investigate these separate cell types in the blood of subjects with asthma and identify which genes are more highly expressed when compared to cells obtained from patients without asthma. We will investigate corticosteroid sensitivity on gene expression in asthma (corticoid naive to corticosteroid resistant asthma). We will also investigate the lung cells (macrophages) from these subjects to identify whether the same or different genes are expressed in these cells.

We will isolate different leukocyte populations from the blood and extract ribonucleic acid (RNA) from these samples. The type and quantity of RNA in these samples is a reflection of the specific genes expressed in these cells. Gene expression is also evaluated by ELISA.This RNA will be sent to Gene Logic in the USA and this company will test these samples to identify which genes have been expressed using Gene Arrays. This technique will examine the expression of all 33,000 human genes in each sample to examine activation of interacting pathways rather than individual genes at a time. Samples will be analysed in the USA and preliminary data shows that there are no problems involving sample transportation or degradation.

Similar experiments will be performed using cells (macrophages) obtained following bronchoalveolar lavage of these subjects. We would aim to examine the responses of cells from two groups of subjects, namely (i) non-asthmatics controls and (ii) asthmatic subjects. The isolated cells will either be immediately solubilized in solutions to purify RNA or we will then use these isolated cells in vitro and following stimulation investigate whether different genes are expressed or at a differential rate in the disease state. We will examine both cells derived from peripheral blood and cells (macrophages) obtained from bronchoalveolar lavage with the aim to determine whether differences attributable to disease can be identified in both circulating cells and those at the site of disease.

This is a preliminary study to determine the profile of inflammatory mediator expression from leukocytes and as such power calculations to determine the number of subjects is not appropriate.

The objective of the study is to identify which genes are specifically expressed in important cells in patients with asthma with a view to identify novel targets for drug therapy.

ELIGIBILITY:
Inclusion Criteria:

Asthmatic Patients

1. Stable asthmatics on beta-2 agonist alone not using more than 4 puffs per day
2. Atopic as defined by positive skin prick tests to at least 2 common aeroallergens
3. PC20 methacholine of < 4 mg /ml
4. Increase in FEV1 > 15% following beta-2 agonist inhalation, either at the time of study or previously documented
5. Age 21-55 years of both sexes (females will be taking adequate contraceptive measures)
6. Non-smokers
7. Normal chest x-ray (CXR) and electrocardiogram (ECG) within the last 6 months.

Healthy Non-Asthmatic Subjects

All normal volunteers will meet the following criteria:

1. Age 21-70 years of both sexes (females will be taking adequate contraceptive measures)
2. No history of respiratory or allergic disease e.g. PC20 methacholine of > 64mg/ml and negative skin prick tests
3. Non-atopic with negative skin prick tests to common aeroallergens
4. Normal baseline spirometry as predicted for age, sex and height.
5. Non-smokers
6. Not taking regular medication
7. No upper respiratory tract infection within the last 6 weeks

Exclusion Criteria:

Subjects will not be included in this study if they meet any of the following exclusion criteria:

1. Clinically significant findings in the medical history or on physical examination other than those of asthma in the asthma group.
2. Lung function FEV1 <30%
3. Pregnant women or mothers who are breastfeeding.
4. Patients who smoke
5. Upper respiratory infection within the last 4 weeks
6. Allergy to local anaesthetic
7. Subjects who are unable to give informed consent.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2003-12; Study Completion 2007-07 (Estimated)

PRIMARY OUTCOMES:
gene expression evaluated using mRNA

SECONDARY OUTCOMES:
corticosteroid sensitivity

CONTACTS AND LOCATIONS:
Overall Officials: Ian M Adcock, PhD, Principal Investigator — NHLI, Imperial College
Locations (1):
- Airway Disease, NHLI, Imperial College, London, United Kingdom